CLINICAL TRIAL: NCT01808508
Title: Obstructive Sleep Apnea and Neurocognitive and Cardiovascular Function in Children With Down Syndrome
Acronym: TRIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-007964
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2015-12

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea Syndrome
Keywords: Down syndrome; Obstructive sleep apnea syndrome; Continuous positive airway pressure; sham or placebo CPAP
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1- Continuous positive airway pressure (CPAP) (Active Comparator): Group 1 will receive therapeutic CPAP for 4 months.
  Interventions: Device: Continuous positive airway pressure
- Group 2-Sham Continuous positive airway pressure (CPAP) (Placebo Comparator): Group 2 are individuals with OSAS who will receive sham or placebo continuous positive airway pressure (CPAP) for 4 months.
  Interventions: Device: Sham or placebo continuous positive airway pressure
- Group 3- No Intervention (No Intervention): Group 3 are individuals with normal breathing during sleep who will not receive any intervention and will be used as a control group.

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure is a machine used with sleep which compresses air delivered via a nasal mask and thus helps stent the airway open.
  Other Names: CPAP
  Arms: Group 1- Continuous positive airway pressure (CPAP)
Device: Sham or placebo continuous positive airway pressure — Sham or placebo CPAP is a machine used instead of therapeutic CPAP. This machine is similar to a therapeutic CPAP machine but has built in leaks and does not deliver pressure. It is not effective in treating OSAS.
  Other Names: Sham or placebo CPAP
  Arms: Group 2-Sham Continuous positive airway pressure (CPAP)

SUMMARY:
Many individuals with Down syndrome (DS) have breathing problems during sleep. This is called obstructive sleep apnea syndrome (OSAS). OSAS is very common in individuals with Down syndrome because of the shape of their face and tongue and because of their low muscle tone. OSAS can cause a lot of health problems including behavioral and learning problems as well as heart problems.

The purpose of this research study is to look at the effects of treating OSAS in individuals with Down syndrome with a machine called Continuous Positive Airway Pressure (CPAP). The investigators want to see if treatment of OSAS improves learning, behavior and heart problems.

DETAILED DESCRIPTION:
All individuals participating in the study will be evaluated for obstructive sleep apnea syndrome (OSAS) with a baseline sleep study. Based on the results of the sleep study,individuals with OSAS will be randomly assigned into two groups. One group will receive continuous positive airway pressure (CPAP) and the other intervention group will receive sham CPAP(placebo) for four months. CPAP is a machine with a mask that fits over the nose, is worn during sleep and helps keep the airway open. Sham CPAP (placebo) is a machine that looks and sounds like a CPAP machine but does not give pressure so it does not treat OSAS. Individuals with normal breathing during the sleep study will not receive a machine, and will serve as controls.

Individuals will also have baseline tests including blood tests, an echocardiogram (pictures of the heart), a walking test and learning tests. After 4 months, the baseline tests will be repeated in all participants. At the end of the study, all individuals with OSAS will get treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 8-20 years
2. Down syndrome (based on the characteristic phenotype)
3. Families provide informed consent and child provides assent

Exclusion Criteria:

1. Subjects and families who do not speak English well enough to undergo psychometric testing.
2. Subjects living in institutions where there is no primary caregiver to participate in the neurocognitive/behavioral battery.
3. Major chronic lung disease such as chronic aspiration.
4. Previous or current CPAP therapy.
5. Participation in a weight loss program.
6. Craniofacial or neuromuscular conditions other than those associated with DS.
7. Untreated hypothyroidism. Participants with normal thyroid function tests will be included in the study.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Marcus, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from The Children's Hospital of Philadelphia Trisomy 21 Program and community support groups.
Pre-assignment Details: 27 subjects were consented, 4 subjects were ineligible before randomization. Subjects with an obstructive apnea hypopnea index (AHI) of at least 5/hr were randomized to CPAP or sham CPAP (Group 1 or 2) for 4 months in a double-blind fashion. Subjects with normal baseline polysomnograms (AHI <1.5/hr) were followed without CPAP (Group 3).
Groups:
- Group 2-Sham Continuous Positive Airway Pressure (CPAP): Group 2 are individuals with OSAS who will receive sham or placebo continuous positive airway pressure (CPAP) for 4 months.
  Sham or placebo continuous positive airway pressure: Sham or placebo CPAP is a machine used instead of therapeutic CPAP.
  This machine is similar to a therapeutic CPAP machine but has built in leaks and does not deliver pressure. It is not effective in treating OSAS.
Period: Overall Study
Arm/Group | Group 1- Continuous Positive Airway Pressure (CPAP) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) | Group 3- No Intervention
Started | 11 | 9 | 3
Completed | 10 | 9 | 3
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 3 - No Intervention: Group 3 are individuals with normal breathing during sleep who will not receive any intervention and will be used as a control group
- Total: Total of all reporting groups
Arm/Group | Group 1- Continuous Positive Airway Pressure (CPAP) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) | Group 3 - No Intervention | Total
Number analyzed (Participants) | 11 | 9 | 3 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.0 [9.0 to 11.5] | 12.0 [9.0 to 15.0] | 12 [10.0 to 13.5] | 10 [9.0 to 14.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 9
  Male | 9 | 4 | 1 | 14
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Epworth Sleepiness Scale From Baseline to End of Study
Description: The primary aim of the study is to assess the relationship between obstructive sleep apnea syndrome (OSAS) and the neurocognitive and behavioral outcomes of individuals with Down syndrome. Sleepiness was assessed using the pediatric version of the Epworth Sleepiness Scale (ESS). The ESS is a self-administered questionnaire with 8 questions. It provides a measure of a person's general level of daytime sleepiness, or average sleep propensity in daily life. The ESS asks people to rate, on a 4-point scale (0, low to 3, high) their usual chances of dozing off or falling asleep in 8 different situations or activities that most people engage in as part of their daily lives. The total ESS score provides an estimate of a general characteristic of each person's average level of sleepiness in daily life (0= no chance of dozing/no daytime sleepiness to 24=high chance of dozing/lots of daytime sleepiness).
Time Frame: 4 Months
Population: 1 OSAS subject randomized to CPAP did not return for follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1- Continuous Positive Airway Pressure (CPAP) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) | Group 3- No Intervention
Number analyzed (Participants) | 10 | 9 | 3
units on a scale | -1 [-4 to 0] | -0.5 [-3 to 0.75] | 1 [0.5 to 3.5]

2. Secondary Outcome: Change in Child Behavior Checklist (CBCL) Total Score From Baseline to 4 Months
Description: The change in behavioral domain was measured by the Child Check Behavior List. The CBCL is a widely used method of identifying problem behavior in children. Problems are identified by a respondent who knows the child well, usually a parent or other care giver. There are 2 versions based on the child's age (CBCL/1½-5 for use children 18 months-5 years; the CBCL/6-18 for children aged 6-18 years). The checklists consists of a number of statements about the child's behavior and responses are recorded on a scale: 0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True. The preschool checklist contains 100 questions and, school-age checklist contains 120 questions. 8 sub-scores (1 for each of 8 syndromes: anxious/depressed, withdrawn depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior and aggressive behavior) are calculated, each ranging from 0 (normal) to 16 (clinical behavior).
Time Frame: 4 Months
Population: 1 OSAS subject randomized to CPAP did not return for follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1- Continuous Positive Airway Pressure (CPAP) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) | Group 3- No Intervention
Number analyzed (Participants) | 10 | 9 | 3
units on a scale | -2 [-4.5 to 0] | 2 [0.75 to 5.25] | 2 [1 to 4.5]

3. Secondary Outcome: Change in the Left Ventricular (LV) Mass Index Score From Baseline to 4 Months
Description: The change in left ventricular mass index score, measured on echocardiography, was used to assess the relationship between obstructive sleep apnea syndrome and cardiovascular function of individuals with Down syndrome. Left ventricular (LV) mass was calculated from M-mode measurements of the LV end-diastolic dimension, the thickness of the interventricular septum and the thickness of the LV posterior wall, and presented as a z-score.
Time Frame: 4 Months
Population: 1 OSAS subject randomized to CPAP did not return for follow-up
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Group 1- Continuous Positive Airway Pressure (CPAP) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) | Group 3- No Intervention
Number analyzed (Participants) | 10 | 9 | 3
z-score | -0.06 [-0.58 to 1.57] | -1.18 [-1.97 to 0.00] | 0.36 [0.12 to 2.71]

4. Secondary Outcome: Change in the Distance Walked on a 6 Minute Walk Test From Baseline to 4 Months
Description: As secondary outcome of the second aim, we will use the distance walked during the 6 minute walk test.
Time Frame: 4 Months
Population: The majority of subjects were unable to follow instructions properly and therefore none could successfully complete the test. Thus the results were not considered to be valid.
Arm/Group | Group 1- Continuous Positive Airway Pressure (CPAP) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) | Group 3- No Intervention
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 Months
Arm/Group | Group 1- Continuous Positive Airway Pressure (CPAP) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) | Group 3- No Intervention
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 1/11 | 2/9 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Continuous Positive Airway Pressure (CPAP) (N=11) | Group 2-Sham Continuous Positive Airway Pressure (CPAP) (N=9) | Group 3- No Intervention (N=3)
Pressure Sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — On forehead from probe used during sleep study
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lyme Disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This preliminary study was limited by the small sample size, and the few children with Down Syndrome but normal breathing during sleep.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes